CLINICAL TRIAL: NCT06696768
Title: Phase I Clinical Trial of CA-4948 (Emavusertib) in Combination With FOLFOX Plus Bevacizumab as Frontline Treatment in Patients With Metastatic Colorectal Cancer
Brief Title: Clinical Trial of an Anti-cancer Drug, CA-4948 (Emavusertib), in Combination With Chemotherapy Treatment (FOLFOX Plus Bevacizumab) in Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-09416; NCI-2024-09416 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10655 (Other: Yale University Cancer Center LAO); 10655 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2024-11-19; First posted 2024-11-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Colorectal Adenocarcinoma; Stage III Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Unresectable Colorectal Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Biopsy; Specimen Handling; CA-4948; Fluorouracil; dehydroftorafur; Leucovorin; Magnetic Resonance Spectroscopy; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (CA-4948, bevacizumab, FOLFOX) (Experimental): Patients receive CA-4948 PO BID on days 1-14 of each cycle, bevacizumab IV over 30-90 minutes on day 1 of each cycle beginning in cycle 1, and oxaliplatin IV over 120 minutes, leucovorin IV over 2 hours, and fluorouracil IV bolus followed by continuous IV infusion over 46 hours on day 1 of each cycle. Cycles repeat every 14 days for up to 2 years in the absence of disease progression or unacceptable toxicity. After treatment for 2 years, patients may continue treatment after discussion with the study chair. Patients also undergo blood sample collection and CT, MRI, or PET/CT throughout the trial. Patients may also undergo tumor biopsy throughout the trial.
  Interventions: Biological: Bevacizumab; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Emavusertib; Drug: Fluorouracil; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Drug: Oxaliplatin; Procedure: Positron Emission Tomography
- Group B (CA-4948, bevacizumab, FOLFOX) (Experimental): Patients receive CA-4948 PO BID on days 1-14 of each cycle, bevacizumab IV over 30-90 minutes on day 1 of each cycle beginning in cycle 2, and oxaliplatin IV over 120 minutes, leucovorin IV over 2 hours, and fluorouracil IV bolus followed by continuous IV infusion over 46 hours on day 1 of each cycle. Cycles repeat every 14 days for up to 2 years in the absence of disease progression or unacceptable toxicity. After treatment for 2 years, patients may continue treatment after discussion with the study chair. Patients also undergo blood sample collection and CT, MRI, or PET/CT throughout the trial. Patients also undergo tumor biopsy throughout the trial.
  Interventions: Biological: Bevacizumab; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Emavusertib; Drug: Fluorouracil; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Drug: Oxaliplatin; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Emavusertib — Given PO
  Other Names: AU 4948; AU-4948; CA 4948; CA-4948; CA4948; Interleukin-1 Receptor-associated Kinase 4 Inhibitor CA-4948; IRAK4 Inhibitor CA-4948
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; Elplat; JM 83; JM-83; JM83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; RP54780; SR 96669; SR-96669; SR96669
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase I trial studies the side effects and best dose of CA-4948 when given together with fluorouracil, leucovorin, oxaliplatin (FOLFOX) plus bevacizumab in treating patients with colorectal cancer that has spread from where it first started (primary site) to other places in the body (metastatic). CA-4948 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. The chemotherapy drugs used in FOLFOX, fluorouracil and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Leucovorin is used with fluorouracil to treat colorectal cancer. Bevacizumab is in a class of medications called anti-angiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to the tumor. This may slow the growth and spread of the tumor. Giving CA-4948 with FOLFOX plus bevacizumab may be safe, tolerable and/or effective in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess dose-limiting toxicities (DLTs) and determine the recommended phase 2 dose (RP2D) of CA-4948 (emavusertib) in combination with leucovorin (folinic acid), fluorouracil, and oxaliplatin (FOLFOX) plus bevacizumab in first-line treatment for patients with advanced or metastatic non-operable colorectal cancer (mCRC).

II. To evaluate the safety and tolerability of the combination of CA-4948 (emavusertib) and FOLFOX plus bevacizumab.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To evaluate ribonucleic acid sequencing (RNAseq) data to examine the impact of interleukin 1 receptor associated kinase 4 (IRAK4) inhibition on downstream signaling in tumor samples.

EXPLORATORY OBJECTIVES:

I. To evaluate pharmacodynamic (PD) effect of CA-4948 (emavusertib) in combination with chemotherapy.

II. To evaluate pharmacokinetics (PKs) of CA-4948 (emavusertib) in combination with chemotherapy.

III. To explore biomarkers and genomic alterations associated with treatment response.

IV. To evaluate if certain gene mutations alone or in combination are associated with response, progression free survival (PFS), and/or overall survival (OS).

OUTLINE: This is a dose-escalation study of CA-4948 in combination with FOLFOX plus bevacizumab followed by a dose-expansion study. Patients are assigned to 1 of 2 groups.

GROUP A: Patients receive CA-4948 orally (PO) twice daily (BID) on days 1-14 of each cycle, bevacizumab intravenously (IV) over 30-90 minutes on day 1 of each cycle beginning in cycle 1, and oxaliplatin IV over 120 minutes, leucovorin calcium (leucovorin) IV over 2 hours, and fluorouracil IV bolus followed by continuous IV infusion over 46 hours on day 1 of each cycle. Cycles repeat every 14 days for up to 2 years in the absence of disease progression or unacceptable toxicity. After treatment for 2 years, patients may continue treatment after discussion with the study chair. Patients also undergo blood sample collection and computed tomography (CT), magnetic resonance imaging (MRI), or positron emission tomography (PET)/CT throughout the trial. Patients may also undergo tumor biopsy throughout the trial.

GROUP B: Patients receive CA-4948 PO BID on days 1-14 of each cycle, bevacizumab IV over 30-90 minutes on day 1 of each cycle beginning in cycle 2, and oxaliplatin IV over 120 minutes, leucovorin IV over 2 hours, and fluorouracil IV bolus followed by continuous IV infusion over 46 hours on day 1 of each cycle. Cycles repeat every 14 days for up to 2 years in the absence of disease progression or unacceptable toxicity. After treatment for 2 years, patients may continue treatment after discussion with the study chair. Patients also undergo blood sample collection and CT, MRI, or PET/CT throughout the trial. Patients also undergo tumor biopsy throughout the trial.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 12 months after end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed colorectal adenocarcinoma
* Patients must have unresectable or metastatic measurable disease on imaging for Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 determination within 28 days of registration
* For patients enrolling to the expansion cohort, lesions must be amenable to research biopsy
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of CA-4948 (emavusertib) and FOLFOX in combination with bevacizumab in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (or Karnofsky ≥ 60%)
* Absolute neutrophil count ≥ 1,500/mcL (within 28 days of registration)
* Platelets ≥ 75,000/mcL (within 28 days of registration)
* Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN) (within 28 days of registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 × institutional ULN; for those with liver metastases, 5 × institutional ULN (within 28 days of registration)
* Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m^2 (within 28 days of registration)
* Creatine phosphokinase (CPK) elevation at screening < grade 2 (CPK ≤ 2.5 x ULN) (within 28 days of registration)
* Patients on a cholesterol lowering statin must be on a stable dose with no dose changes within 3 weeks prior to study start
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible, after discussion with the principal investigator (PI) or medical monitor, if the treating physician determines that immediate CNS-specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* Patients must be able to take oral medications
* The effects of CA-4948 (emavusertib) on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Women of childbearing potential must continue contraception for 9 months following the last dose of study drugs. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Males treated or enrolled on this protocol and involved with women of childbearing potential must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 6 months following the last dose of study drugs
* Patients must have the ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients with high-frequency microsatellite instability (MSI-H) or deficient deoxyribonucleic acid (DNA) mismatch repair (dMMR) colorectal cancer at pre-enrollment screening
* Patients with prolonged QT interval by Fridericia's correction formula (QTcF) (> 450ms) on screening electrocardiogram (ECG)
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1), with the exception of alopecia
* Patients who are receiving any other investigational agents
* Patients who have received prior treatment with any chemotherapy (either in the adjuvant or metastatic setting), including FOLFOX, fluorouracil/leucovorin/irinotecan (FOLFIRI), folinic acid/fluorouracil/oxaliplatin/irinotecan (FOLFOXIRI), or antiangiogenic agents such as bevacizumab and similar agents, are not eligible for this study
* Patients with a known dihydropyrimidine dehydrogenase deficiency
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to CA-4948 (emavusertib) or other agents used in the study
* Patients with a gastrointestinal (GI) condition that could impair absorption of CA-4948 (emavusertib) or cause an inability to ingest CA-4948 (emavusertib)
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because CA-4948 (emavusertib) is a blood-brain barrier penetrant with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CA-4948 (emavusertib), breastfeeding should be discontinued if the mother is treated with CA-4948 (emavusertib). These potential risks may also apply to other agents used in this study. Women of childbearing potential must have a negative pregnancy test within 7 days of study entry
* Patients with a history of allogeneic organ or stem cell transplantation
* Patients with significant active bleeding or those in whom the treating physician believes bevacizumab would not be safe or appropriate
* Patients who have had palliative radiation to bone metastases within 2 weeks prior to day 1 of the study treatment
* Patients who have had a major surgical procedure within 4 weeks prior to day 1 of the study treatment
* Patients with hypertension not controlled by antihypertensive medication
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 14 days prior to randomization; however,

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea; or chronic daily treatment with corticosteroids with a dose of ≤ 10 mg/day methylprednisolone equivalent) may be enrolled
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Severe infections within 28 days prior to registration, including but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia. This includes receipt of oral or IV antibiotics within 14 days prior to registration. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) | Up to 2 cycles (Cycle length = 14 days)
  DLT will be based on the first 2 cycles (28 days) of emavusertib.
Incidence of treatment-emergent adverse events | Up to 2 cycles (Cycle length = 14 days)
  The adverse events will be recorded by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.

SECONDARY OUTCOMES:
Incidence of adverse events | Baseline to 30 days after last dose of study drug
  Adverse events, graded according to the National Cancer Institute CTCAE v5 for each cohort, will be analyzed using descriptive statistics.
Overall response rate | From the start of treatment until disease progression/recurrence, assessed up to 12 months after end of treatment
  Defined as the percentage of patients who achieve complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1.
Progression free survival | From first dose to the earlier date of assessment of progression or death by any cause in the absence of progression, assessed up to 12 months after end of treatment
  Will be assessed using RECIST v1.1.
Overall survival | From the date of first dose to the date of death by any cause, assessed up to 12 months after end of treatment
Disease control rate | Up to 12 months after end of treatment
  Defined as the percentage of patients who achieve a best response of CR, PR, or stable disease (SD) per RECIST v1.1 at any time during their treatment. A determination of SD requires that the first restaging imaging scan be performed after 4 cycles of treatment (8 weeks from start of treatment +/- 7 days).
Molecular profiling | At baseline, between cycle (C) 1 day (D) 10 and C1D14, and disease progression
  Molecular profiling by next generation sequencing will be done to assess the impact of IRAK4 inhibition on downstream signaling in tumor samples.

OTHER OUTCOMES:
Pharmacodynamic (PD) biomarkers | At baseline, between C1D10 and C1D14, and disease progression
  PD biomarkers including p-IRAK4, p-p65, p-ERK by immunohistochemistry (IHC) to determine the effect of IRAK4 inhibition by emavusertib before and after treatment will be analyzed using two-way analysis of variation (ANOVA) followed by post-doc pairwise comparison test.
Pharmacokinetic (PK) parameters | C1D1, 0.5, 1, 2, 4, 6, and 8 hours post-dose on C2D1, C3D1
  Emavusertib steady-state PK parameters will be estimated, specifically maximum concentration, area under the concentration-time curve, and apparent clearance using non-compartmental methods. PK parameters will be reported descriptively for exploratory comparison with historical data. Advanced population PK methods may be employed at a later stage to assess the link between drug exposure and biological effects and efficacy.
Immune profiling | At baseline, day 1 of each cycle, and 30 days after last dose of study drug
  Multiplex IHC will be used to assess T cell infiltrates, activation, and exhaustion, as well as myeloid and dendritic cell panels before and after treatment. This will be analyzed using a Wilcoxon signed-rank test.
Systemic immunity in circulation | On C1D1, C2D1, and C3D1 and at progression
  This analysis will be performed using blood samples collected on the same day (+/- 3 days) as tumor biopsy. Will employ a 36-parameter cytometry by time-of-flight panel designed for adaptive and innate immune cells. Changes in each marker before and after treatment will be analyzed using two-way ANOVA followed by post-hoc pairwise comparison test.
Multiplex cytokine/chemokine analysis | On C1D1, C2D1, C3D1, and disease progression
  Multiplex cytokine/chemokine analysis IL-1α/β, IL-6, IL-8 and IFN-γ, CCL2, CXCL1, CXDL2 that may be diminished by IRAK4 inhibition. This analysis will be performed using blood samples. A customized panel of 25 analytes will be used to profile all biomarkers and correlate with patients' clinical outcomes. Changes in each marker before and after treatment will be analyzed using two-way ANOVA followed by post-hoc pairwise comparison test.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna V Ulahannan, Principal Investigator — Yale University Cancer Center LAO
Locations (13):
- United States (13):
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Hospital East, Shiloh, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm